CLINICAL TRIAL: NCT01413620
Title: Vitamin E Supplementation in Burn Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: University of Texas (Other); Oregon State University (Other)
Responsible Party: Principal Investigator, Jong O. Lee, Assistant Professor of Surgery and Faculty Surgeon, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VitE2011
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Burn Injury
Keywords: Vitamin E; Burn; Oxidation; Lung Dysfunction; Fatty Liver; Lipid Peroxidation
MeSH Terms: conditions — Burns; Fatty Liver | interventions — alpha-Tocopherol; Vitamin E

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin E Treated (Experimental)
  Interventions: Drug: dl-alpha-tocopheryl acetate
- Untreated (No Intervention)

INTERVENTIONS:
Drug: dl-alpha-tocopheryl acetate — Ages 6 months-1 year will receive 75 IU/day of dl-alpha-tocopheryl acetate, while ages 2-5 years will receive 150 IU/day. Ages 6-8 will receive 300 IU/day, while ages 9-13 will receive 600 IU/day, ages 14-17 will receive 800 IU/day, and ages 18-70 will receive 1200 IU/day. Vitamin E will be administered in a liquid or pill form. The dose of aqueous vitamin E (Aqueous Vitamin E Oral Drops, Silarx, No. 54838-0005-30, Spring Valley, NY) will be given orally. When/If the patient is able to eat independently, the dose of vitamin E may be given in a pill form (Novatol 5-57, No. 410217, Archer Daniels Midland Company, Decatur, IL). Depending on the subject's group, the supplement of vitamin E either will be given on days 1-15 of the study or days 16-30 of the study.
  Other Names: Vitamin E; Aqueous Vitamin E Oral Drops, Silarx, No. 54838-0005-30
  Arms: Vitamin E Treated

SUMMARY:
Burned patients because of their increased oxidative stress have severely depleted vitamin E, which is a dietary antioxidant. Oxidative stress is responsible for much of the pathophysiology seen in burned patients, which leads to acute and chronic morbidity and mortality, in addition to a decrease in their quality of life. Oral vitamin E will be used to reverse the oxidative stress of burn injury and, in the process, decrease the secondary consequences of thermal trauma. This proposal will demonstrate the benefit of maintaining adequate vitamin E status.

DETAILED DESCRIPTION:
We have previously demonstrated that thermal injury depletes plasma vitamin E in pediatric burn patients. However, plasma changes reflect short-term vitamin E changes, whereas adipose tissue alpha-tocopherol concentrations reflect long-term vitamin E status. We reported last year that burn injury depleted vitamin E stores in adipose tissue in children by nearly half within one month following injury. Our long-term goal is to improve the quality of life of burn patients by preventing pulmonary and hepatic dysfunction that may occur from vitamin E depletion. The objectives of this application are to a) attenuate alpha-tocopherol depletion in burned patients by vitamin E supplementation, b) prevent or reverse oxidative stress in these patients, and c) collect pilot data on the effect of vitamin E supplementation on lung and liver function. Our central hypothesis is that the administration of high doses of alpha-tocopherol will prevent or restore levels of vitamin E in adipose tissue and reverse the oxidative state in burned patients. The rationale of the proposed studies is that in severe cases of vitamin E depletion, oxidative stress, fatty liver and lung dysfunction have all been reported in our patients. We will administer vitamin E supplements (300-1200 IU RRR-alpha-tocopherol) to burn subjects (n= 20 per group, 6-70 years, ≥20% total body surface burns) for fifteen days. The subjects will be randomly assigned into two groups: an early treatment group who will receive vitamin E for days 1-15 of the study, and a delayed treatment group who will receive vitamin E for days 16-30 of the study. Both groups will be studied for a total of thirty days. We will test the following aims: Aim 1: determine the degree that supplemental Vitamin E will attenuate alpha-tocopherol depletion. Aim 2: determine if supplemental Vitamin E reduces markers of oxidative stress in burned patients. Aim 3: collect preliminary data to establish the relationship between oxidative stress and pulmonary pathophysiology and fatty liver after burn injury. We will measure plasma and adipose tissue alpha-tocopherol and urinary and plasma markers of oxidative stress, prior to supplementation and then weekly. The proposed research is innovative because the oxidative stress of burn injury causes a severe depletion of an essential nutrient, vitamin E. Supplementation of vitamin E is a novel concept that may mitigate the complications of burns, including lung injury, fatty liver and peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 months - 85 years
* >20% TBSA burn

Exclusion Criteria:

* Bleeding disorders
* Positive hepatitis or HIV screens
* Pregnancy (women)

Ages: 6 Months to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2017-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Alpha-Tocopherol in Plasma, Adipose (also: Lung, Skin, Muscle, Liver in the case of Death) | 30 Days
Gamma-Tocopherol in Plasma, Adipose (also: Lung, Skin, Muscle, Liver in the case of Death) | 30 Days
Vitamin E Metabolites in Plasma, Urine | 30 Days
Malondialdehyde in Plasma, Urine (also: Lung, Skin, Muscle in the case of Death) | 30 Days
Isoprostanes in Plasma, Urine (also: Lung, Skin, Muscle in the case of Death) | 30 Days
Lipid Panel in Plasma and Triglyceride Concentration | 30 Days
Liver Ultrasound | 30 Days
Pulmonary Function Study Variables | 30 Days
Cardiopulmonary Stress Test | 30 Days

SECONDARY OUTCOMES:
Open Body Surface Area and Wound Healing | 30 Days
Weight | 30 Days
Basal Metabolic Rate | 30 Days
Diet History and Food Intake | 30 Days
Fluid Balance | 30 Days
Incidence of Acute Respiratory Distress Syndrome (ARDS) | 30 Days
Incidence of Pneumonia | 30 Days
Incidence of Atelectasis | 30 Days
Ventilator Variables (Compliance, Resistance, Work of Breathing, Number of Days Ventilated) | 30 Days
Pulmonary Status Variables (Spirometry, Blood Gas, Diffusion Constant, Pulmonary Capillary Surface Area) | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Jong O Lee, MD, Principal Investigator — University of Texas Medical Branch, Shriners Hospitals for Children; Hal K Hawkins, MD, PhD, Study Director — University of Texas Medical Branch, Shriners Hospitals for Children; Linda E Sousse, PhD, MBA, Study Director — University of Texas Medical Branch, Shriners Hospitals for Children; Daniel L Traber, PhD, Study Director — University of Texas Medical Branch, Shriners Hospitals for Children; Maret G Traber, PhD, Study Director — Oregon State University; David N Herndon, M.D., Study Director — University of Texas Medical Branch, Shriners Hospitals for Children; Celeste C Finnerty, Ph.D., Study Director — University of Texas Medical Branch, Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No